CLINICAL TRIAL: NCT05644288
Title: Impact of the HELPeN Telecare Program on Social Isolation and Loneliness in Community-dwelling Elders: Randomized Control Trial
Brief Title: Impact of the HELPeN Program on Social Isolation in Community-dwelling Elders (HELPeN)
Acronym: HELPeN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MARIA RUZAFA MARTINEZ (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundación Poncemar (Unknown)
Responsible Party: Sponsor-Investigator, MARIA RUZAFA MARTINEZ, Associate Professor. Faculty of Nursing. University of Murcia, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PI21/00984
Record Dates: First submitted 2022-11-26; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Loneliness; Isolation, Social
Keywords: Loneliness; Isolation, Social; Elderly people; Telenursing; Volunteers
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: Two-arm parallel stratified randomized clinical trial with 12 months duration performing measurements at time 0, 3, 6, 9 and 12 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data will be collected by three team members who will make a telephone call to the study participants and record the study variables on four occasions throughout the study. They will be blinded, i.e., they will have no information about the major. Also, the data analyst will not know to which group each subject belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The proposed intervention is a telephonic telenursing program aimed at managing social isolation in the elderly, the HELPeN (Help eNursing) program.
  The operational part of the intervention will be carried out by volunteers nursing students from the University of Murcia enrolled in the academic years 2020-2023. To ensure homogeneity in the intervention carried out by the volunteers they will receive a 15-hour training oriented to ensure the acquisition of essential communication skills for the implementation of the intervention and to know the specific interventions of support and counseling for the elderly in social isolation.
  Interventions: Other: Help eNursing
- Control group (No Intervention): No intervention will be performed in the control group and the subjects will be contacted on the same dates as the intervention group for data collection.

INTERVENTIONS:
Other: Help eNursing — The proposed intervention is a telephonic telenursing program aimed at managing social isolation in the elderly, the HELPeN (Help eNursing) program.
  The operational part of the intervention will be carried out by volunteers nursing students from the University of Murcia enrolled in the academic years 2020-2023. To ensure homogeneity in the intervention carried out by the volunteers they will receive a 15-hour training oriented to ensure the acquisition of essential communication skills for the implementation of the intervention and to know the specific interventions of support and counseling for the elderly in social isolation.
  Over the 36 weeks of the HELPeN Program, each volunteer is expected to provide intervention to 2 seniors, making 1 call per week to each subject lasting approximately 30 minutes. Students will perform physical and psychosocial assessments of the elders and create individualized care plans based on each subject's needs.
  Arms: Intervention group

SUMMARY:
The main objective is to determine the effectiveness of the HELPeN Program, a 12-month telephone telenursing program for community-dwelling elderly in social isolation, evaluating the main changes in levels of social isolation, loneliness, quality of life, mental health status (depression), sleep and functional capacity, as well as changes in care management (demand for services and consumption of drugs).

Methodology Two-arm parallel stratified randomized clinical trial with 12 months duration performing measurements at time 0, 3, 6, 6, 9 and 12 months.

Participating subjects will be selected by nursing professionals from users of Area 3 of Health of the Region of Murcia over 65 years old, residing in the community and with a Social Isolation score <32 (Low perceived social support with DUFSS). Randomization will be performed after stratification according to whether the subjects live alone or accompanied, with a 1:1 ratio. Given an alpha level of 0.05, an anticipated effect size of 1.58, beta power equal to 1, 42 subjects are required in each group.

The intervention consists of a telephonic telenursing program HELPeN (Help eNursing) to be carried out in collaboration with the Poncemar Volunteer Bank.

The control group will not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* score < 32 (Low perceived social support with the DUFSS scale)
* Residence in the community

Exclusion Criteria:

* Severe cognitive impairment (8-10 errors on the Pfeiffer test)
* Non Spanish speakers
* Failure to consent to the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Loneliness | 9 months
  Name of the measurement: Loneliness
  Definition: Loneliness is the result of a cognitive evaluation where there are discrepancies between the social relationships that people desire and those that they really have.
  Measuremente tool: UCLA Loniness Scale. Developed by psychologist Daniel Russell (1996), the UCLA Loneliness Scale (Version 3) is a 20-item measure that assesses how often a person feels disconnected from others.
  Unit of measure: Indicence of loneliness
Social isolation | 9 months
  Name of the measurement: Social isolation
  Definition: Disengagement from social relationships, connections with institutions or community involvement.
  Measurement tool: DUKE-UNC Functional Social Support questionnaire(DUFSS). A 14-item, self-administered, multidimensional, functional social support questionnaire.
  Unit of measure: Incidence of social isolation

SECONDARY OUTCOMES:
Phisycal function | 9 months
  Name of the measurement: Phisycal function
  Definition: The level of functional independence of patients with neuromuscular and musculoskeletal pathologies
  Measurement tool: Barthel Index for Activities of Daily Living. Scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.
  Unit of measure: % of subjects "able to live independently"; "minimally dependent"; "partially dependent"; "very dependent"; "total dependece"
Depression | 9 months
  Name of the measurment: Depression
  Definition: Depression is a common but serious mood disorder. It causes severe symptoms that affect how you feel, think, and handle daily activities, such as sleeping, eating, or working.
  Measurement tool: Geriatric Depression Scale (GDS). The original scale consists of 30 dichotomous items (Yes/No), and direct scoring, between 0 and 30.
  Unit of measure: Incidence of depression and mean punctuation in the GDS scale
Mental status | 9 months
  Name of the measurement: Mental status
  Definition:
  Measuremente tool: Short portable mental status questionnaire (SPMSQ) (Pfeiffer's test). It is a brief questionnaire composed of ten questions that measure the degree of cognitive impairment. Evaluates cognitive impairment for the purpose of screening for dementia. Heteroapplied.
  Unit of measure: Incidence of cognitive impairment and % of subject with "intact intellectual functioning"; "intact intellectual functioning"; "moderate intellectual impairment" and "severe intellectual impairment"
Anxiety | 9 months
  Name of the measuremente: Anxiety
  Definition: Generalized anxiety disorder (GAD) include clearly excessive, uncontrollable, and often irrational anxiety and worry of a duration of at least 6 months
  Measuremente tool: 7-item Generalized Anxiety Disorder Scale (GAD-7). It is a 7 items self-report scale designed to identify probable cases of GAD.
  Unit of measure: % of subjects with "minimal anxiety"; "mild anxiety"; "severe anxiety"
Health Related Quality of life | 9 months
  Name of the measurement: Health Related Quality of life
  Definition: It encompass those aspects of overall quality of life that can be clearly shown to affect health-either physical or mental
  Measuremente tool: European Quality of Life-5 Dimension (EQ-5D). It can be used at the individual level to monitor a patient's health status over time. The EQ-5D instrument consists of 2 parts - the EQ-5D descriptive system and the Visual Analog Scale (VAS). The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. In the VAS the individual scores his or her health between two extremes, 0 and 100, the worst and the best state of health imaginable.
  Unit of measure: % of subjects reporting health problems by level in each dimension. Mean punctuation of the VAS scale.
Health assistance | 9 months
  Name of the measurement: Health assistance
  Definition: Health care provided to a patient including: hospitalization, face-to-face or telephone consultation, home care, visit to emergency department and the professional providing the care.
  Measuremente tool: these information will be collected from electronic record of the patients
  Unit of measure:% of subjects requiring health assistance: hospitalization, face-to-face or telephone consultation, home care, visit to emergency department and the professional providing the care.
Drugs | 9 months
  Name of the measurement: Consumption of drugs
  Definition: the prescription or increase in daily dosage, according to the anatomical-therapeutic classification (ATC) of the WHO, of the following drugs will be recorded: Psycholeptics, Psychoanaleptics, Analgesics, Muscle relaxants and Other drugs.
  Measuremente tool: prescriptions will be collected from electronic record of the patients
  Unit of measure: % of subjects taking Psycholeptics, Psychoanaleptics, Analgesics, Muscle relaxants and Other drugs.

CONTACTS AND LOCATIONS:
Overall Officials: César Leal-Costa, RN, PhD, Principal Investigator — Universidad de Murcia; María Ruzafa-Martínez, RN, PhD, Principal Investigator — Universidad de Murcia
Locations (1):
- Healthcare Area III. Region of Murcia, Lorca, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided